CLINICAL TRIAL: NCT01823562
Title: Dietary Fruit Bioactives and Prostate Cancer
Brief Title: Aborption and Metabolism of Lyophilized Black Raspberry Food Products in Men With Prostate Cancer Undergoing Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-12125; NCI-2013-00326 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
Keywords: Lyophilized Black Raspberry; Prostate Cancer; Surgery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm I (regular diet) (Active Comparator): Patients follow a regular diet for 4-6 weeks and then undergo prostatectomy.
  Interventions: Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (low polyphenol diet) (Active Comparator): Patients follow a low polyphenol diet for 4-6 weeks and then undergo prostatectomy.
  Interventions: Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm III (low ellagitannin diet) (Active Comparator): Patients follow a low ellagitannin diet for 4-6 weeks and then undergo prostatectomy.
  Interventions: Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm IV (lower-dose lyophilized black raspberry gummy) (Experimental): Patients follow a low ellagitannin diet and receive lower-dose black raspberry gummy PO daily for 4-6 weeks and then undergo prostatectomy.
  Interventions: Drug: lyophilized black raspberry confection; Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm V (higher-dose black raspberry gummy) (Experimental): Patients follow a low ellagitannin diet and receive higher-dose black raspberry gummy PO daily for 4-6 weeks and then undergo prostatectomy.
  Interventions: Drug: lyophilized black raspberry confection; Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm VI (lower-dose black raspberry confection) (Experimental): Patients follow a low ellagitannin diet and receive lower-dose black raspberry confection PO daily for 4-6 weeks and then undergo prostatectomy.
  Interventions: Drug: lyophilized black raspberry confection; Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm VII (higher-dose black raspberry confection) (Experimental): Patients follow a low ellagitannin diet and receive higher-dose black raspberry confection PO daily for 4-6 weeks and then undergo prostatectomy.
  Interventions: Drug: lyophilized black raspberry confection; Other: laboratory biomarker analysis; Dietary Supplement: dietary intervention; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Drug: lyophilized black raspberry confection — Given PO
  Other Names: LBR confection
  Arms: Arm IV (lower-dose lyophilized black raspberry gummy); Arm V (higher-dose black raspberry gummy); Arm VI (lower-dose black raspberry confection); Arm VII (higher-dose black raspberry confection)
Other: laboratory biomarker analysis — Correlative studies
Dietary Supplement: dietary intervention — Follow a low polyphenol diet
  Other Names: Dietary Modification; intervention, dietary
  Arms: Arm II (low polyphenol diet)
Dietary Supplement: dietary intervention — Follow a low ellagitannin diet
  Other Names: Dietary Modification; intervention, dietary
  Arms: Arm III (low ellagitannin diet); Arm IV (lower-dose lyophilized black raspberry gummy); Arm V (higher-dose black raspberry gummy); Arm VI (lower-dose black raspberry confection); Arm VII (higher-dose black raspberry confection)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This Phase I/Ib trial is studying the absorption and metabolism of phytochemicals found in black raspberries in men undergoing surgery for prostate cancer. This knowledge will help us design future chemoprevention studies and assist in making future dietary recommendations for men at high risk for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a dose-escalation study to determine safety and compliance of varying lyophilized black raspberry (LBR) delivery vehicles (a gummy confection and a nectar) at two different doses.

SECONDARY OBJECTIVES:

I. To precisely quantify changes in the content and distribution of black raspberry phytochemicals and their metabolites in the blood and urine and correlate these concentrations with prostate tissue phytochemicals.

II. Measure the ability of black raspberry gummy confection and nectar in altering hormonal patterns (lower insulin-like growth factor-1 [IGF-I], higher insulin-like growth factor-binding protein 3 [IGF-BP3], lower androgens) consistent with reduced prostate carcinogenesis and in parallel with an enhanced capacity to quench reactive oxygen.

III. Investigate histopathologic, immunologic, and molecular biomarkers associated with prostate carcinogenesis that may serve as surrogate endpoint biomarkers and provide information regarding their ability to be modulated by black raspberries.

IV. Determine if consumption of black raspberries alters molecular markers in the human prostate including: (a) neuroendocrine markers such as IGF-I and IGF-BP3, (b) signal transduction markers such as phosphatase and tensin homologue (PTEN) and phospho-AKT, and (c) angiogenesis regulators such as (vascular epithelial growth factor (VEGF).

V. Collect and store plasma and peripheral blood mononuclear cells (PBMCs) from each patient to assess systemic markers of inflammation and immune response.

OUTLINE: This is a dose-escalation study of lyophilized black raspberry gummy confection and nectar. Patients are assigned to 1 of 7 treatment arms.

ARM I: Patients follow a regular diet for 4-6 weeks and then undergo prostatectomy.

ARM II: Patients follow a low polyphenol diet for 4-6 weeks and then undergo prostatectomy.

ARM III: Patients follow a low ellagitannin diet for 4-6 weeks and then undergo prostatectomy.

ARM IV: Patients follow a low ellagitannin diet and receive lower-dose black raspberry gummy orally (PO) daily for 4-6 weeks and then undergo prostatectomy.

ARM V: Patients follow a low ellagitannin diet and receive higher-dose black raspberry gummy PO daily for 4-6 weeks and then undergo prostatectomy.

ARM VI: Patients follow a low ellagitannin diet and receive lower-dose black raspberry nectar PO daily for 4-6 weeks and then undergo prostatectomy.

ARM VII: Patients follow a low ellagitannin diet and receive higher-dose black raspberry nectar PO daily for 4-6 weeks and then undergo prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy proven carcinoma of the prostate
* Have chosen a radical prostatectomy for treatment of their disease after the medical team has presented all possible treatment options
* Not be receiving neoadjuvant hormonal or chemotherapy (other clinical trials)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Not currently taking berry dietary supplements, or "alternative" products (Acai berry, pomegranate, black raspberry, Optiberry, Juice Plus)
* Have BUN/Cr (blood urea nitrogen and serum creatinine) within normal limits
* Have liver enzymes within normal limits
* Have complete blood count (CBC) within normal limits
* Have prothrombin time/partial thromboplastin time (PT/PTT/INR) within normal limits
* Voluntarily agree to participate and sign an informed consent document
* Agree to have prostate biopsy blocks provided to the study for evaluation
* Agree to consume a standardized vitamin and mineral supplement and avoid other nutrition, dietary, or alternative medications/supplements for the duration of the study
* Agree to follow a controlled polyphenolic and/ or ellagitannin diet

Exclusion Criteria:

* Have an active malignancy other than prostate cancer that requires therapy
* Have a prostate biopsy with less than 5% cancer involvement
* Have a history of traumatic or surgical castration
* Have a history of pituitary hormone diseases that currently require supplemental hormonal administration (thyroid hormones, adrenocorticotropic hormone [ACTH], growth hormone) or other endocrine disorders requiring hormone administration with the exception of diabetes and osteoporosis
* Are taking certain medications; no concurrent finasteride (Proscar) or other hormonal agents for chemoprevention/treatment of benign prostate hyperplasia (BPH); utilizing prescription medications for urinary outlet obstructive symptoms will not be permitted; the use of non-prescription substances to improve urinary tract symptoms will not be permitted (i.e. Saw Palmetto, other herbal, alternative products)
* Have a known allergy to black raspberries, corn, and wheat products or those who have never consumed any of these products
* Have active metabolic or digestive illnesses such as malabsorptive disorders (Crohn's, Celiac disease, irritable bowel syndrome [IBS]), renal insufficiency, hepatic insufficiency, cachexia, or short bowel syndrome
* Have significant loss of gastrointestinal organs due to surgery, except for appendix
* Have altered immunity such as autoimmune disorders, cancer, anemia, hemophilia, and blood dyscrasias
* Have noticeable open lesions in the oral cavity, sores that have not healed for more than 2 months or have a history of leukoplakia, tumors of the buccal cavity, throat, and lips
* Have difficulty swallowing (dysphagia), pain with swallowing (odynophagia), salivary gland dysfunction, or xerostomia (dry mouth)
* Are taking medications that inhibit clotting (warfarin sodium) or using prescribed oral rinses (Peridex)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days after completion of study treatment
Compliance determined by consumption of at least 80% of black raspberries (BRB) and positive tests for urinary berry metabolites | Up to 6 weeks
  A cohort will be considered compliant if the group mean consumption of the intervention product is at least 80%.

SECONDARY OUTCOMES:
Presence of black raspberry metabolites in the urine collected 24 hours before surgery | Up to 6 weeks
  Analyzed on the log scale using a repeated measures linear model to judge the effect of treatment group in terms of fold-differences from baseline while controlling for body mass index (BMI) and age. Confidence intervals for dichotomous variables will be made using exact methods and confidence intervals for rank correlations between quantitative variables will be made using Fisher's transformation.
Changes in PSA or PSA doubling time | Up to 6 weeks
  Analyzed on the log scale using a repeated measures linear model to judge the effect of treatment group in terms of fold-differences from baseline while controlling for BMI and age. Confidence intervals for dichotomous variables will be made using exact methods and confidence intervals for rank correlations between quantitative variables will be made using Fisher's transformation.
Black Raspberry metabolites levels in the prostate tissue removed at surgery | Up to 6 weeks
  Confidence intervals for dichotomous variables will be made using exact methods and confidence intervals for rank correlations between quantitative variables will be made using Fisher's transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu